CLINICAL TRIAL: NCT05423639
Title: The Influence of Lateral Pressure on Sectional Matrix in Optimizing Proximal Contact Tightness in Class II Resin Composite Restoration
Brief Title: Influence of Lateral Pressure on Sectional Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Salem Sayed Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29301030104462
Record Dates: First submitted 2022-05-05; First posted 2022-06-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Class II Dental Caries

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group 1 (Experimental): Testing Palodent sectional matrix system only when placing Class II resin composite restorations is to increase proximal contact tightness.
  Interventions: Device: palodent
- Intervention group 2 (Active Comparator): A pre-contoured instrument called Optra contact (Ivoclar, Vivadent) will be used with group 2. For testing palodent matrix systems with Optracontact when placing Class II resin composite restorations is to increase proximal contact tightness with adjacent teeth when compared with group 1.
  Interventions: Device: palodent; Device: optracontact

INTERVENTIONS:
Device: palodent — innovative sectional matrix system with Nickel-Titanium rings, anatomically shaped matrix bands and adaptive self-guiding wedges that provides predictable, tight contacts and restorations that accurately replicate the natural tooth anatomy.
  Other Names: sectional matrix system
Device: optracontact — The instrument is used to achieve large and tight proximal contacts in posterior teeth.
  Other Names: Molar Instrument - Ivoclar Vivadent; Bifurcated Tip Instrument
  Arms: Intervention group 2

SUMMARY:
The aim of this study was evaluating the clinical effectiveness of the hand instrument in conjunction with sectional matrix when applying lateral forces at the contact area during curing to achieve large and tight proximal contacts in posterior teeth.

DETAILED DESCRIPTION:
Dental caries is considered as one of the most prevalent oral infections. Initiation of dental caries is a mufti-factorial process, its risk factors includes high loads of cariogenic bacteria, increased frequency of sugar intake, insufficient exposure to fluoride and reduced salivary flow. Other factors that may influence the occurrence of caries include poor oral hygiene and socio-economic status.

Inter-proximal caries lesions develop between the contacting proximal surfaces of two adjacent teeth. Massive evolution took place in restorative techniques, composite resin materials, cavity designs and armamentarium in the past few decades. As well as drastic solutions for earlier problems of composite resins such as bonding to dentin, wear resistance, postoperative sensitivity and polymerization shrinkage. Despite all the progress noted in that area, still achieving proximal contact tightness in Class II resin composite restorations is considered one of the biggest challenges facing clinicians Proximal contact tightness is a physiological dynamic entity of multifactorial origin that is largely affected by tooth type, location, time of day, patient position, mastication and restorative procedures Failure to obtain proper proximal contact area will influence stability of dental arch and transmission of forces along long axis of teeth during mastication. Traumatic masticatory forces can lead to various problems like; rotation and displacement of the teeth, lifting forces on the teeth, deflective occlusal contacts and food impactions that would result in trauma, pain, inflammation and bleeding of the periodontium. The contact must be neither open nor too tight.

Aim of this study was evaluating the clinical effectiveness of the Optra Contact in conjunction with sectional matrix when applying lateral forces at the contact area during curing to achieve large and tight proximal contacts in posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients having posterior class II carious lesions were included
* Absence of pain from the tooth to be restored
* Good general health
* Age range:18-50 years
* Fully erupted occluding teeth

Exclusion Criteria:

* Diastema between posterior teeth
* Presence of fixed partial dentures
* Severe periodontal diseases Tooth mobility Non vital teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Contact tightness Device used: Dental floss Scoring unit US Public Health Service | Proximal contact tightness was measured after 6 months
  Clinical Performance Proximal contact Modified USPHS Ryge criteria

CONTACTS AND LOCATIONS:
Overall Officials: sara SA sayed, master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt